CLINICAL TRIAL: NCT01801891
Title: Surface NeuroMuscular Electrical Stimulation in the Treatment of Chronic Venous Leg Ulcers: A Randomised Controlled Trial of the "VASGARD" Device
Brief Title: Surface NeuroMuscular Electrical Stimulation in the Treatment of Chronic Venous Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Professor Stewart Walsh (Other)
Responsible Party: Sponsor-Investigator, Professor Stewart Walsh, Professor Stewart Walsh, Mid Western Regional Hospital, Ireland
Organization: Mid Western Regional Hospital, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VASGARD2013
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Venous Disease
Keywords: Venous ulceration; Leg ulcers; Venous haemodynamics; Surface neuromuscular electrical stimulation; SNMES
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer | interventions — Compression Bandages

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Patients randomised to the control group will, in addition to their routine compression bandaging, be given muscle stimulators for home use and instructed to apply 3x 30 minute sessions of comfortable electrical stimulation daily for 12 weeks. The stimulators given to the control group will be set to provide minimal stimulation resulting in no visible muscular contraction.
  Interventions: Other: Compression bandaging
- VASGARD stimulator (Experimental): Patients randomised to this group, in addition to their routine treatment with compression bandaging, will be given muscle stimulators for home use and instructed to apply 3x 30 minute sessions of comfortable electrical stimulation daily for 12 weeks. The intervention group stimulators will be capable of causing muscular contraction with a maximum force ranging from 30-40% of voluntary contractions.
  Interventions: Device: VASGARD stimulator; Other: Compression bandaging

INTERVENTIONS:
Device: VASGARD stimulator — The VASGARD device is a 2 channel muscle stimulator system designed for increasing venous blood flow. Controlled electrical stimuli are delivered to the patient through adhesive gel electrodes placed over the motor points of muscles on the lower leg. This elicits artificial muscular contractions which in turn increases lower limb venous haemodynamics.
  Other Names: SNMES
  Arms: VASGARD stimulator
Other: Compression bandaging — Compression bandaging systems apply graduated external pressure to the lower limb to promote venous return to the heart reducing venous hypertension and thereby facilitate venous ulcer healing.
  Other Names: Graduated compression bandaging

SUMMARY:
This study aims to determine if the use of surface neuromuscular electrical stimulation, applied to various motor points on the lower limb to elicit muscle contraction when combined with compression bandaging accelerates the rate of venous leg ulcer healing.

DETAILED DESCRIPTION:
With an increasingly ageing population the incidence of venous ulceration is likely to rise. The negative impact of leg ulceration on patients' quality of life and on healthcare costs is well recognised. Increased prevalence combined with poor reported healing rates and high incidence of ulcer recurrence makes the development of a new treatment which could accelerate healing rates beyond that currently achieved using compression bandaging most desirable. Surface neuromuscular electrical stimulation in combination with compression bandaging may provide such a treatment.

Surface neuromuscular electrical stimulation (SNMES) is the application of an electrical stimulus to motor points in the body using electrodes placed on the surface of the skin to elicit a muscular contraction. It has been shown that SNMES of the calf muscles, when used in conjunction with compression therapy, provides improved venous flow velocities over compression therapy alone. Furthermore, the week-long effect of SNMES and compression therapy on healthy participants was found to be well tolerated by all participants and resulted in increases in stimulated venous flow and muscle strength. A combined SNMES and compression treatment protocol which stimulates peripheral venous blood flow may help to alleviate harmful venous pressures in venous leg ulcer patients and provide some degree of strengthening of the calf muscles, thus helping to accelerate the healing rates of venous ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent venous leg ulcer.
* Ankle-brachial pressure index > 0.8
* Ulcer size between 1 and 200 cm2
* Patient suitable for full compression bandaging

Exclusion Criteria:

* History of symptomatic heart disease.
* Pregnancy
* Presence of implants in the lower leg or a pacemaker
* History of a neurological disorder
* Presence of any contraindications for the use of compression stockings such as severe arterial disease i.e. Ankle brachial pressure index (ABPI) <0.8
* Presence of cognitive difficulties which may prevent the patient or his/her carer from using the stimulator appropriately.
* Patients unable to provide informed consent
* Patients receiving dialysis
* Patients receiving steroids
* Patients receiving methotrexate
* Ulcer located in the area of electrode placement
* Patients in reduced compression bandaging system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reduction in venous ulcer size | 12 weeks
  Reduction in relative ulcer size (area) for each patient over time, standardised to an initial size of 1, will be measured weekly.

SECONDARY OUTCOMES:
Acceptability of surface neuromuscular electrical stimulation | 12 weeks
  Patient and healthcare provider perceptions of the acceptability, efficacy and tolerability of the device will be evaluated through a series of semi-structured interviews

OTHER OUTCOMES:
Changes in skin condition related to the application of Vasgard surface neuromuscular electrical stimulator as a measure of safety and tolerability. | 12 weeks
  The safety issues associated with using electrical stimulation on this patient group under compression bandaging will be evaluated. The following safety points will be evaluated at each visit.
  1. Appearance of the skin under the electrodes (intact / reddened / broken)
  2. Appearance of skin surrounding the electrodes (intact / reddened /broken)
  3. Appearance of skin under the electrodes leads (intact / reddened / broken

CONTACTS AND LOCATIONS:
Overall Officials: Pierce A Grace, MCh FRCSI, Principal Investigator — HSE
Locations (2):
- Ireland (2):
  - Department of Electronic Engineering, National University Ireland Galway, Galway
  - MidWestern Regional Hospital, Limerick